CLINICAL TRIAL: NCT07217548
Title: Solving Stigma Through POV Simulation: Enhancing Pharmacist Empathy-based Practices With Sickle Cell Disease Patients
Acronym: point of view
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Howard University (Other); Fairleigh Dickinson University (Other); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Nicholas Denton, Senior Lecturer, Ohio State University
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: UM1TR004548 (NIH); UM1TR004548 (NIH)
Record Dates: First submitted 2025-10-03; First posted 2025-10-16 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Stigma
Keywords: pharmacists; PharmD students
MeSH Terms: conditions — Social Stigma

STUDY DESIGN:
Intervention Model Description: Participants will be invited to complete the intervention arm or control arm, followed by assessment.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be unaware of the other arm (POV simulation vs control intervention) and outcome assessors of empathy-based practice will be unaware of which arm participants belong to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- POV simulation (Experimental): Participating pharmacists in the experimental arm will receive an email invitation to complete a 16-item pre-survey around opioid use misconceptions before completing the point of view simulation activity. 10 days after participants complete the simulation they will be invited to complete the opioid misconception survey again as a post-learning intervention assessment. 6 months after participants complete the simulation, their practice site will be visited by a sickle cell disease patient evaluator who will refill their opioid medication with the pharmacist and then complete an 11-item evaluation survey on the pharmacist's empathy-based pharmacy practices.
  Interventions: Behavioral: point of view simulation
- Control (Sham Comparator): Participating pharmacists in the sham arm will receive an email invitation to complete a 16-item pre-survey around opioid use misconceptions before completing an unrelated hematology educational activity. 10 days after participants complete the simulation they will be invited to complete the opioid misconception survey again as a post-learning intervention assessment. 6 months after participants complete the simulation, their practice site will be visited by a sickle cell disease patient evaluator who will refill their opioid medication with the pharmacist and then complete an 11-item evaluation survey on the pharmacist's empathy-based pharmacy practices.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: point of view simulation — In POV simulations, participants actively engage with a patient looking to fill an opioid script at a community pharmacy setting through the point of view of the pharmacist. Using a "choose your own adventure" branch chain format, our research team has already drafted interaction pathways where participants can respond to the patient with empathy-based practice, act on a common misconception around chronic opioid use, or mislabel the patient as drug seeking. After 3-4 interaction branches, the participants reach a decision to fill the opioid script, deny it, or some variation of delaying the script being filled. The POV simulation then replays the participant's choices back to them from the patient's point of view, revealing that the SCD patient was in genuine pain and engaging participant's empathy as they rewatch their microaggressive and mislabeled drug seeker choices through the patient's POV.
  Arms: POV simulation
Behavioral: Control — Participants will watch a hematology educational video unrelated to pain management
  Arms: Control

SUMMARY:
Why This Research Matters (Significance)

1 in 5 of the 50+ million people with chronic pain in the U.S. face stigma when using opioids, especially women and racial minorities. This stigma often comes from pharmacy staff treating chronic pain patients as drug seekers, who then refuse to fill the patient's script, and leave the patient in severe pain. The team has found that having pharmacists watch testimonial videos of sickle cell patients sharing their pain management struggles can help reduce these misconceptions. However, using point of view simulations could be even more effective in fostering empathy among pharmacists. The goal is to create an educational simulation that helps pharmacists better understand and manage pain in sickle cell patients, ultimately improving their care.

What Makes This Research Unique (Innovation) Traditional methods to address biases in healthcare include watching patient testimonials or using expensive actors to play a standardized patient interaction to health professionals. This innovative point of view simulations engage participants' empathy more effectively by playing back what participants told the patient from the patient's point of view and are more accessible by having participants interact with the simulation on the computer any time and any place, rather than organizing a paid actor to visit the hospital. With advancements in artificial intelligence, we can create interactive simulations where virtual patients respond dynamically to questions, making the experience more realistic and impactful.

How Will the Researchers Conduct the Research (Approach)

The researchers will test if point of view simulations can reduce misconceptions among healthcare professionals and improve pain management for sickle cell patients. Here's the plan:

1. Create and Implement the Simulation: Use it as part of the training for pharmacy and hospital staff, as well as nursing and pharmacy students.
2. Survey Participants: Before and after the simulation, participants will take a survey to measure their misconceptions about opioid use.
3. Follow-Up: Six months later, researchers will survey the participants' patients and their managers to see if there's been an improvement in the empathetic care the participants provided.

DETAILED DESCRIPTION:
1. SIGNIFICANCE An unintended translational science challenge of the opioid epidemic is that >20% of the 50+ million chronic pain patients in the US alone face opioid use stigma from pharmacy staff that has left them in debilitating pain.1 Within this cohort of stigmatized patients there's a higher portion of women and girls that have been harmed by misogynistic stereotypes of "hysteric" and "oversensitive" women exaggerating their pain, resulting in pharmacists questioning the legitimacy of their pain more than male chronic pain patients.2,3 Likewise, there's also a higher portion of Black chronic patients undertreated in their pain as racial stereotypes of Black Americans as "criminals" and "drug addicts" due to racial trauma inflected during the US War on Drugs result in Black patients being disproportionately mislabeled as drug-seeking.4 Health professional training often perpetuates misconceptions like "melanin makes skin thicker" and "white skin has more free nerve endings" that also contribute to implicit bias against giving Black patients the same level of pain management as their white counterparts.5 Woman sickle cell disease (SCD) patients are particularly vulnerable to being mislabeled as drug-seeking due to misogynistic and racist stereotyping intersectionality while managing debilitating pain from relatively invisible vaso-occlusion crisis that necessitates chronic opioid use and eventual breakthrough pain as opioid tolerance develops.6,7

   While the project team has previously demonstrated that SCD patient testimonial videos partially alleviates common opioid misconceptions shared by pharmacists, the limited translation of knowledge from educational interventions to noticeable change in pharmacists' practice remains a critical knowledge gap. While tasking pharmacists to passively watch patient testimonials sharing their struggles in pain management did result in significant decreases in agreement scores to misconceptions like "opioids are always dangerous when used long term" or "a patient can receive great care without being treated for pain", baseline agreement was already very low to discriminatory statements like "race has a negligible impact on the perception of a patient's drug habits" despite continued discrimination in pharmacy practice. This disconnect between learners' knowledge of health disparities and self-awareness of deficiencies in their practice is likely due to the implicit nature of bias where microaggressions against patients persist unnoticed by the healthcare professional.8

   The proposed research aligns with the translational science definition through practical application of our previous research and others' scientific discoveries toward creating innovative point-of-view (POV) simulations through a collaborative approach including an interdisciplinary research team alongside SCD community partners, with broad applicability across not just SCD patient biases but other patient-healthcare professional interactions where microaggressions negatively impact health outcomes. The central theme is to create a freely distributed and empathetically impactful educational simulation that results in better health outcomes for SCD patients. Primary goals are to recruit SCD community partners in the quick and efficient production of the POV simulation, to broadly implement the simulation into continuing education workshops and courses throughout our collaborative network, and to rigorously and ethically assess whether the POV simulation decreases pharmacists' agreement toward opioid use misconceptions and whether SCD patients observe quality improvements in their pharmacy's empathy-based care practices.
2. INNOVATION The predominate clinical education practices to address implicit basis include participant's passively watching patient testimonials or hiring cost-prohibitory standardized patients; our research team includes pioneers in POV simulation technologies that have the potential to drive engaging and accessible educational interventions against healthcare professional biases against SCD patients. In POV simulations, participants actively engage with a patient looking to fill an opioid script at a community pharmacy setting through the point of view of the pharmacist. Using a "choose your own adventure" branch chain format, the research team has already drafted interaction pathways where participants can respond to the patient with empathy-based practice, act on a common misconception around chronic opioid use, or mislabel the patient as drug seeking. After 3-4 interaction branches, the participants reach a decision to fill the opioid script, deny it, or some variation of delaying the script being filled. The POV simulation then replays the participant's choices back to them from the patient's point of view, revealing that the SCD patient was in genuine pain and engaging participant's empathy as they rewatch their microaggressive and mislabeled drug seeker choices through the patient's POV. In addition to leveraging empathy-based learning, POV simulations can be engaged asynchronously online and repeated as many times as participants want, making POV simulations much more accessible to health professionals than training and scheduling a standardized patient actor to roleplay the simulation.9 With advancements in AI technology, there's also potential to enhance the authenticity and therefore impact of the interaction by incorporating chatbot-like AI patients that dynamically respond to participants interview questions rather than following a set script for a case study.
3. APPROACH To test the hypothesis that POV simulations can alleviate misconceptions in health professionals and improve pain management outcomes in SCD patients, the research team first aims to create a POV SCD patient simulation that is engages empathy in participants and is authentic to the SCD patient experience. The research team of SCD hematology, palliative care, health disparity, and education technology experts have already drafted branching interaction scripts that include authentic misconceptions, microaggressions, and empathy-based care responses observed in pharmacy practices. SCD patient and advocates from community partners at the Faith Thomas Foundation engage in the translational science process by consulting on the authenticity of the simulation.

   The next aim is to assess whether the POV simulation alleviates the misconceptions around opioid use that are most detrimental toward chronic pain patients by implementing the learning intervention within the research team's various institutions that include pharmacy/ER staff and nursing/PharmD students who serve >2,000 SCD patients. Staff participants will be incentivized with continuing education credit while student participants will receive a course assessment grade to take our experimentally validated, 16-item opioid stigma misconceptions Likert survey right before completing the POV simulation and again 10 days afterwards along with a reflection on any specific microaggressions or misconceptions that participants realized they had around chronic opioid use. Community partners will likewise consult on the survey design to validate the impact of the survey questions on SCD opioid use stigma.

   The final aim will be to determine whether the POV simulation caused noticeable change in healthcare participants' empathy-based care practices and SCD patient health outcomes by surveying SCD patient simulated patients. Six months after completing the POV simulation, participants' and non-participant controls' SCD patients will also be invited to complete a 12-item expert-validated Likert survey on their healthcare professional's empathetic care practices and microaggressions along with a free response question on their overall satisfaction in their pain management outcomes to assess for impactful changes in SCD patient care (Fig. 3). Survey data will be collected via Qualtrics and stored on a secure drive in compliance with OSU's data storage and sharing policies. Multivariate analysis of survey participants' agreement scores will control for differences in their practice site, demographics (gender, race/ethnicity, age, etc.), and any close relationships they have with SCD or opioid use disorder when determining whether POV simulations alleviated health professional participants' misconceptions and improved SCD patient outcomes.
4. HEALTH EQUITY The community partner, the Faith Thomas Foundation, has agreed to recruit SCD patients and advocates that will be engaged in every phase of the translational process in the project design. To reduce any potential biases or misconceptions the POV simulation producers and actors might have about SCD patients, reviewing the simulation scripts and guiding the actors to make sure the SCD patient experience is authentically represented in the simulation. Likewise, SCD consultants would be able to assist in ethically recruiting a representative population of SCD patients from the research team's combined network of >2,000 patients to provide authentic assessment of their health outcomes rather than relying solely on self-reported observations from the health professionals. By creating an engaging, empathetic, and accessible educational intervention, this project has the potential to expand beyond the >2,000 SCD patients within the research team's network toward reducing health disparities and debilitating pain for the 10+ million chronic pain patients that encounter stigma for their opioid use.

ELIGIBILITY:
Inclusion Criteria:

* Practicing healthcare professional OR student in a healthcare professional program
* Ability to fill opioid prescriptions

Exclusion Criteria:

* Not currently practicing or rotating in a clinical setting that fills opioid prescriptions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Agreement/disagreement toward opioid use misconceptions | Baseline and 10 days post-treatment
  An experimentally validated, 16-item opioid stigma misconceptions survey right before starting the POV simulation and again 10 days afterwards with the aim to assess alleviation of misconceptions most impactful to chronic pain patients such as sickle cell disease patients.
Frequency of empathy-based care practices when filling opioid prescriptions | 3 months post-treatment
  Three months after completing the POV simulation, sickle cell patients on the research team will also be invited to complete a 12-item expert-validated survey on the participants' empathetic care with the aim to assess impacts of the POV simulation on patient care.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas L Denton, PhD, Principal Investigator — Ohio State University College of Pharmacy
Locations (1):
- Ohio State University College of Pharmacy, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
As part of the informed consent process, the research team promises participants that their individual deidentified data will not be shared with other researchers.

REFERENCES:
- [Background] Sinha CB, Bakshi N, Ross D, Krishnamurti L. Management of Chronic Pain in Adults Living With Sickle Cell Disease in the Era of the Opioid Epidemic: A Qualitative Study. JAMA Netw Open. 2019 May 3;2(5):e194410. doi: 10.1001/jamanetworkopen.2019.4410. PMID 31125105
- [Background] Carroll CP. Opioid treatment for acute and chronic pain in patients with sickle cell disease. Neurosci Lett. 2020 Jan 1;714:134534. doi: 10.1016/j.neulet.2019.134534. Epub 2019 Oct 5. PMID 31593753
- [Background] Samulowitz A, Gremyr I, Eriksson E, Hensing G. "Brave Men" and "Emotional Women": A Theory-Guided Literature Review on Gender Bias in Health Care and Gendered Norms towards Patients with Chronic Pain. Pain Res Manag. 2018 Feb 25;2018:6358624. doi: 10.1155/2018/6358624. eCollection 2018. PMID 29682130
- [Background] Grant AD, Miller MM, Anastas TM, Quinn P, Lok B, Hirsh AT. Opioid-related risk perceptions in chronic pain: influence of patient gender and previous misuse behaviors. Pain. 2022 Apr 1;163(4):711-718. doi: 10.1097/j.pain.0000000000002412. PMID 34285152